CLINICAL TRIAL: NCT04248959
Title: Prehabilitation to Improve Cancer Surgery Outcomes in AYA Patients With Extremity Sarcomas (PICaSO-ES): A Proof-of-Concept Trial
Brief Title: Prehabilitation to Improve Cancer Surgery Outcomes in AYA Patients With Extremity Sarcomas
Acronym: PICaSO-ES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: MOUNT SINAI HOSPITAL (Other)
Responsible Party: Principal Investigator, Daniel Santa Mina, Clinician Investigator, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-5901; 18-0226 (Other: Toronto Academic Health Sciences Network)
Record Dates: First submitted 2020-01-22; First posted 2020-01-30 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Sarcoma,Soft Tissue; Osteosarcoma
Keywords: Preoperative Care; Exercise Therapy; Prehabilitation; Extremity Sarcoma; Adolescents and Young Adults
MeSH Terms: conditions — Sarcoma; Osteosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multimodal Prehabilitation (Experimental): Facility and home-based multimodal prehabilitation (aerobic exercise training, resistance exercise training, nutrition support, stress management and mindfulness training)
  Interventions: Behavioral: Multimodal prehabilitation

INTERVENTIONS:
Behavioral: Multimodal prehabilitation — Multimodal Prehabilitation
  * Aerobic exercise
    * Home-based, high-intensity interval training (HIIT), 2 days/week
    * Home-based, moderate-intensity continuous training (MICT), 2-3 days/week
  * Resistance exercise
    * Home-based, moderate-intensity resistance training, 2-3 d/wk, all major muscle groups (working around tumour-related deficits), 8-10 exercises, 12-15 repetitions, resistance bands and body weight based
  * Nutrition
    * Protein intake 1.2-1.5 g/kg body weight/day in compliance with European Society for Clinical Nutrition and Metabolism (ESPEN) guidelines
  * Stress management
    * Daily mindfulness practice, 20 min/session, guided by audio file created at Mount Sinai Hospital

SUMMARY:
The purpose of this study was to evaluate the feasibility of a multimodal prehabilitation intervention intended to optimize postoperative recovery in adolescents and young adults (AYAs) diagnosed with soft tissue and bone-based sarcomas of the upper and lower extremities (extremity sarcomas; ES).

DETAILED DESCRIPTION:
Objectives:

This objective of this study was to investigate the feasibility of multimodal prehabilitation for adolescents and young adults (AYAs) diagnosed with soft tissue and bone-based sarcomas of the upper and lower extremities (extremity sarcomas; ES) and explore its effects on measurements of health-related quality of life, physical function, length of hospital stays, and post-operative complications. Specific aims of the study included:

* To determine the feasibility of conducting a larger phase II investigation of HIIT-based multimodal prehabilitation according to three primary criteria, including (i) recruiting >=50% of otherwise eligible patients (OEP; i.e., patients meeting all eligibility criteria), (ii) no patient experiences a testing-related or an intervention-related serious adverse event (SAE), and (iii) patients achieve an exercise intervention adherence rate of >=70%.
* To further determine the feasibility of conducting a larger phase II investigation of HIIT-based multimodal prehabilitation according to the secondary feasibility criteria.
* To explore the preliminary effects of prehabilitation on measures of short-term perioperative outcomes including health-related quality of life, physical function, length of hospital stays, and post-operative complications.

Methods:

A single-arm, proof-of-concept trial design was informed by the ORBIT model of behavioural treatment development. Mixed methods were employed to obtain relevant context for investigating the feasibility of multimodal prehabilitation in newly diagnosed AYAs with ES within the circumstances of the COVID-19 pandemic.

Participants underwent virtual multimodal prehabilitation before undergoing major extremity sarcoma surgery. This program encompassed personalized exercise, nutrition, and stress management support delivered by a registered kinesiologist, registered dietitian, and clinical psychologist, respectively. The interventions were designed to enhance physical and psychological resilience to stress, with the objective of improving recovery outcomes and mitigating the risk of adverse events.

Feasibility (e.g., recruitment, safety, tolerability), physical function, and patient-reported outcomes were measured at baseline (T0), immediately preoperatively (T1), and one month postoperatively (T2).

Feasibility data and field notes were collected by the research coordinators (during recruitment and postoperative follow-up) and by the study lead / research assistants during the intervention period. A postoperative interview explored experiences with prehabilitation into explore the feasibility and practical considerations of virtual prehabilitation for adolescents and young adults with extremity sarcomas.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years and <40 years of age at diagnosis
* Fluent in English
* Able to comply with study and follow-up procedures contained within the consent form
* Pathologically or radiologically confirmed diagnosis of a soft-tissue or osteosarcoma of the upper or lower extremities
* Soft-tissue or osteosarcoma must be considered operable
* Patients of all weight bearing states will be eligible
* Expected LOS ≥ 5 days as calculated by the validated American College of Surgeons Surgical Risk Calculator
* >14 days between time of randomization and time of expected surgery
* Patient written, informed consent obtained according to ICH GCP guidelines and local regulations
* Medical clearance to participate in the study from either the primary treating surgeon (JW, PF) or oncologist (AG)

Exclusion Criteria:

* Planned resection of bony pelvis or major lower extremity neurovascular structures
* Significant comorbidity including any of the following:

  * Canadian Cardiovascular Society class III/IV coronary disease
  * New York Heart Association class III/IV congestive heart failure
  * Neurologic or musculoskeletal disorder prohibiting exercise
  * Major neuropsychiatric disorder
* High-risk or presence of pathological fracture

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Patient recruitment rate (feasibility target: >=50% of eligible participants) | Initiation through end of study recruitment at 12 months
  Defined as the percent of consenting patients based on the total number of otherwise eligible patients (OEP; patients meeting all study eligibility criteria) approached
Testing- and intervention-related serious adverse events (feasibility target: none) | Initiation through end of pre-operative testing
  Defined as the number and frequency of testing- and intervention-related serious adverse events (SAEs) according to the Common Terminology Criteria for Adverse Events
Patient exercise adherence (feasibility target: >=70% of prescribed) | Initiation through end of study intervention period
  Defined as relative dose intensity as the percent of total dose of exercise performed relative to the total planned dose prescribed and quantified according to metabolic equivalents

SECONDARY OUTCOMES:
Patient identification rate (feasibility target: >=50% of OEP) | Initiation through end of study recruitmentat 12 months
  Defined as the average number of OEP identified each month
Baseline assessment rate (feasibility target: >=90% of consenting participants) | Initiation through end of study recruitment at 12 months
  Defined as the percent of consenting patients who successfully complete baseline assessments based on the total number of consenting patients
Intervention window (feasibility target: >=21 days) | Initiation through end of study intervention period
  Defined as the average elapsed time (in days) between diagnosis and extremity sarcoma surgery
Testing- and intervention-related non-serious adverse events (feasibility target: <20% of sessions) | Initiation through end of pre-operative testing
  Defined as the number and frequency of testing- and intervention-related non-serious adverse events (nSAEs) according to the Common Terminology Criteria for Adverse Events
Testing performance (feasibility target: >=95% completion of tests) | Initiation through end of pre-operative testing
  Defined as percent completion physical testing at baseline and follow-up
Testing modality adaptations (descriptive) | Initiation through end of pre-operative testing
  Defined as the percent of all tests which are adapted for functional or safety reasons
Training modality adaptations (descriptive) | Initiation through end of study intervention period
  Defined as the percent of all exercise sessions which are adapted for functional or safety reasons
Permanent treatment discontinuation (feasibility target: <=15% of participants) | Initiation through end of study intervention period
  Defined as the percent of patients who discontinue intervention participation prior to the planned end of the intervention period
Treatment interruption (feasibility target: <=15% of participants) | Initiation through end of study intervention period
  Defined as the percent of patients who miss ≥3 consecutive sessions within the intervention period
Dose modification (feasibility target: <=25% of participants) | Initiation through end of study intervention period
  Defined as the percent of exercise sessions requiring a dose reduction during training (i.e., intensity or duration) relative to the total number of sessions completed. Total number of exercise sessions with a reduction in intensity or a reduction in duration will be combined into the numerator when calculating the percentage of affected sessions.
Early session termination (feasibility target: <=25% of participants) | Initiation through end of study intervention period
  Defined as the percent of exercise sessions requiring unplanned early termination
Pretreatment intensity modification (feasibility target: <=25% of participants) | Initiation through end of study intervention period
  Defined as the percent of sessions which required pre-exercise modification of the target exercise intensity due to a pre-exercise screening indication (e.g., fatigue, pain)
Physical prehabilitation compliance (feasibility target: >=70% of prescribed) | Initiation through end of study intervention period
  Defined as the percent of exercise sessions completed based on the total number of sessions prescribed
Mindfulness prehabilitation compliance (feasibility target: >=70% of prescribed) | Initiation through end of study intervention period
  Defined as the percent of psychological sessions completed based on the total number of sessions prescribed
Attrition (feasibility target: <=20% loss to follow-up) | Study initiation through end of 1 month postoperative (T2)
  Defined as the percent loss to follow-up (not completing follow-up assessments), individually and overall

OTHER OUTCOMES:
Global health score | Baseline (T0), preoperative (T1), 1 month postoperative (T2)
  Primary exploratory outcome: European Organization for the Research and Treatment of Cancer (EORTC) QLC-C30
Postoperative complications | 1 month postoperative (T2)
  Postoperative complication severity and frequency defined according to the Common Terminology Criteria for Adverse Events.
Length of stay | 1 month postoperative (T2)
  Average postoperative hospitalization period
Functional capacity | Baseline (T0), preoperative (T1)
  Total distance traveled during six-minute walk test
Physical activity behavior (subjective) | Baseline (T0), preoperative (T1), 1 month postoperative (T2)
  Godin Leisure-time Exercise Questionnaire
Health-related quality of life | Baseline (T0), preoperative (T1), 1 month postoperative (T2)
  EQ-5D; All 5 items are rated on a 1 to 3 scale with higher numbers reflecting worse outcomes.
Symptom burden | Baseline (T0), preoperative (T1), 1 month postoperative (T2)
  Edmonton Symptom Assessment Scale (ESAS); All 10 items are rated on a 0 to 10 scale with higher numbers reflecting worse outcomes.
Anxiety and depression | Baseline (T0), preoperative (T1), 1 month postoperative (T2)
  Hospital Anxiety and Depression Scale (HADS); All 14 items are rated on a 0 to 3 scale with higher numbers reflecting worse outcomes.
Fatigue | Baseline (T0), preoperative (T1), 1 month postoperative (T2)
  Functional Assessment of Chronic Illness Therapy-Fatigue scale (FACIT-F); All 13 items are rated on a 0 to 4 scale with higher numbers reflecting worse outcomes.
Impact on work | Baseline (T0), preoperative (T1), 1 month postoperative (T2)
  Work Limitations Questionnaire
Social support | Baseline (T0), preoperative (T1), 1 month postoperative (T2)
  Medical Outcomes Study Social Support Scale (SF-20); All item scores transformed into 0 to 100 scales with higher scores reflecting better outcomes.
Relationships | Baseline (T0), preoperative (T1), 1 month postoperative (T2)
  Experiences in Close Relationships scale (ECR); All 36 items rated on a 1 to 7 scale with higher scores reflecting worse outcomes.
Extremity function | Baseline (T0), preoperative (T1), 1 month postoperative (T2)
  Toronto Extremity Salvage Score (upper or lower)
Disease burden | Baseline (T0), preoperative (T1), 1 month postoperative (T2)
  Musculoskeletal Tumor Society score

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Santa Mina, PhD, Principal Investigator — University of Toronto; University Health Network
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No